CLINICAL TRIAL: NCT06912048
Title: Understanding Individual Variability in Neuronal Signal Transmission to Target Organs in Health and Disease
Acronym: CPB_Atropine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Martin Heni, Prof. Dr. med. Martin Heni, University of Ulm
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 467/2024; 101125605 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Autonomic Function
Keywords: parasympathetic transmission; autonomic nervous system; brain periphery crosstalk; metabolism; insulin sensitivity; insulin secretion; endogenous glucose production; sex differences; high risk population
MeSH Terms: conditions — Insulin Resistance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atropine Infusion (Experimental): 5 µg x kg fat free mass-1 x h-1
  Interventions: Other: Oral glucose tolerance test with double-tracer dilution and atropine infusion
- Saline infusion (Placebo Comparator)
  Interventions: Other: Oral glucose tolerance test with double-tracer dilution and saline infusion (placebo)

INTERVENTIONS:
Other: Oral glucose tolerance test with double-tracer dilution and atropine infusion — Subjects will undergo a 75 g oGTT (180 min) combined with a double tracer dilution. The double-tracer dilution technique will be used to quantify endogenous glucose production, glucose appearance and disappearance rate. [6,6-2H]glucose will be infused for a total of 300 minutes, while the infusion will start 120 minutes prior the oGTT and will last until the end of the oGTT. Atropine infusion will be administered 20 minutes before the start of the oGTT. The drink consumed at time point 0 min contains 75 gram glucose, enriched with [U-13C6]-glucose.
  Arms: Atropine Infusion
Other: Oral glucose tolerance test with double-tracer dilution and saline infusion (placebo) — Subjects will undergo a 75 g oGTT (180 min) combined with a double tracer dilution. The double-tracer dilution technique will be used to quantify endogenous glucose production, glucose appearance and disappearance rate. [6,6-2H]glucose will be infused for a total of 300 minutes, while the infusion will start 120 minutes prior the oGTT and will last until the end of the oGTT. Saline infusion will be administered 20 minutes before the start of the oGTT. The drink consumed at time point 0 min contains 75 gram glucose, enriched with [U-13C6]-glucose.
  Arms: Saline infusion

SUMMARY:
The goal of this clinical trial is to evaluate the influence of parasympathetic transmission from the brain to different metabolic organs. This transmission can be blocked with the muscarinic antagonist atropine.

Participants will undergo an oral glucose tolerance test combined with a double tracer dilution technique either with atropine infusion or placebo.

Healthy individuals and high-risk individuals will be compared to identify possible changes in signaling in high-risk groups. In addition, men and women will be included to take into account possible sex differences.

DETAILED DESCRIPTION:
This research project aims to investigate to what extent the parasympathetic nervous system is responsible for the transmission of signals from the brain to peripheral organs. Furthermore, the study will investigate sex differences and differences between healthy and high-risk individuals on brain-derived coordination of postprandial signaling for metabolic control.

Therefore, parasympathetic blockade will be introduced by atropine infusion (on one day) versus saline infusion as placebo (on another day) in a randomized fashion. For safety reasons, only the participants will be blinded. Infusion will start 20 minutes before a 75 gram oral glucose tolerance test (oGTT) and last until the end of the 2h oGTT. The oGTT will introduce a postprandial state. Additionally, 1000 mg Paracetamol will be added to the solution to study gastric emptying.

This approach will be combined with a double-tracer dilution technique. Labeled glucose ([6,6-2H]glucose) will be infused 120 minutes before and during the oGTT (120 min) and will be used to address endogenous glucose production. The glucose drink from the oGTT will be enriched with [U-13C6]glucose to compute the glucose appearance rate (Ra). Basal endogenous glucose production will be calculated as well as post-load endogenous glucose production and rates of glucose disappearances (Rd).

ELIGIBILITY:
Inclusion Criteria:

* Age: at least 18
* BMI: 20 - 24.9 kg/m2 (for the healthy groups) or more than 28 kg/m2 (for the overweight groups)
* For women: Hormonal contraception with a single-phase preparation (e.g. Nuvaring)
* Understanding and voluntarily signing an informed consent form prior to study-related examinations

Exclusion Criteria:

* Drug and/or alcohol abuse
* smoking
* Taking medication that affects blood sugar or addresses the central and/or autonomic nervous system (e.g. anti-epileptic drugs, beta blockers, dopamine agonists, antidepressants). Taking antihistamines.
* Pre-existing cardiac conditions
* Neurological pre-existing conditions
* Known cardiac arrhythmia
* Known allergies to ingredients, e.g. paracetamol and atropine
* Known narrow-angle glaucoma
* Known hyperthyroidism
* Known diseases of the urinary tract or prostate
* Pregnancy or breastfeeding
* At screening: Hb < 12 g/dl for women and Hb < 14 g/dl for men
* No consent to be informed about incidentally discovered pathological findings
* Any (clinical) condition which, in the opinion of the physician, could jeopardize the safety of the
* or would jeopardize the scientific success.
* Liver dysfunction
* Renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on glucose tolerance assessed as area under the glucose curve (0-120 minutes) and glucose levels at timepoint 120 minutes during the 75 g oral glucose tolerance test.
Insulin Sensitivity | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on insulin sensitivity assessed from glucose and insulin measurements during the 75 g oral glucose tolerance test.
Insulin Secretion | 180 minutes
  Effect of parasympathetic blockade with atropine versus placebo on insulin secretion assessed from glucose and insulin/C-peptide measurements during the 75 g oral glucose tolerance test.

SECONDARY OUTCOMES:
Lipolysis | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on the suppression of lipolysis during a 75 g oral glucose tolerance test.
Gastric emptying | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on gastric emptying during the 75 g oral glucose tolerance test.
Amino Acid Metabolism | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on amino acid metabolism assessed by amino acid measurements during the 75 g oral glucose tolerance test.
Bile acid metabolism | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on bile acid metabolism assessed by bile acid measurements during the 75 g oral glucose tolerance test.
Substrate oxidation | 230 Minutes
  Effect of parasympathetic blockade with atropine versus placebo on substrate oxidation assessed by indirect calorimetry at timepoints -110 Minutes, 30 Minutes, 60 Minutes and 120 Minutes during the 75 g oral glucose tolerance test.
Incretin secretion | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on incretin secretion during the 75 g oral glucose tolerance test.
Sex differences | 180 minutes
  Explore sex differences in the effect of parasympathetic blockade with atropine versus placebo in the mentioned outcome measures.
Autonomic nervous system | 180 minutes
  Effect of parasympathetic blockade with atropine versus placebo on the autonomic nervous system assessed by heart rate variability during the 75 g oral glucose tolerance test.
Blood coagulation parameters | 120 Minutes
  Influence of of parasympathetic blockade with atropine versus placebo on blood coagulation parameters. This is assessed through global coagulation tests and single coagulation factors.

OTHER OUTCOMES:
Circulating peptides | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on circulating proteins/peptides during the 75 g oral glucose tolerance test.
Lipids and lipoproteins | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on lipids and lipoproteins assessed by lipid measurements during the 75 g oral glucose tolerance test.
Metabolites | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on circulating metabolites during the 75 g oral glucose tolerance test.
Immune cell composition | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on immune cell composition assessed by flow cytometry during the 75 g oral glucose tolerance test.
Insulin clearance | 120 minutes
  Effect of parasympathetic blockade with atropine versus placebo on insulin clearance assessed from insulin and C-peptide measurements during the 75 g oral glucose tolerance test.
Metabolic flexibility | 180 minutes
  Effect of parasympathetic blockade with atropine versus placebo on metabolic flexibility assessed by the change in respiratory quotient during the 75 g oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, MD, Principal Investigator — Ulm University Hopital
Locations (1):
- Ulm University Hospital, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No